CLINICAL TRIAL: NCT00654628
Title: Begin With The Right Patients With Dual-Inhibition Action Therapy Through Vytorin for Newly Diagnosed Dyslipidemia Patients
Brief Title: Begin With The Right Patients With Dual-Inhibition Action Therapy Through Vytorin for Newly Diagnosed Dyslipidemia Patients (0653A-172)(COMPLETED)
Acronym: BRAVO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0653A-172; 2008_010
Record Dates: First submitted 2008-04-02; First posted 2008-04-08 (Estimated); Results first posted 2010-08-26 (Estimated); Last update posted 2024-05-22 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Ezetimibe, Simvastatin Drug Combination

ARMS (1):
- 1 (Experimental): Patients with intermediate or high risk dyslipidemia will be enrolled to receive treatment with Vytorin 10/20 (ezetimibe 10 mg /simvastatin20 mg) tablet once daily consecutively for 6 weeks
  Interventions: Drug: ezetimibe (+) simvastatin

INTERVENTIONS:
Drug: ezetimibe (+) simvastatin — Vytorin 10/20 (ezetimibe 10 mg /simvastatin20 mg) tablet once daily consecutively for 6 weeks.
  Other Names: Vytorin®; MK653A

SUMMARY:
The purpose of this study is to determine the safety and tolerability of ezetimibe/simvastatin in patients newly diagnosed with dyslipidemia.

ELIGIBILITY:
Inclusion Criteria:

* Male Or Female Patient, 20 Through 79 Years Of Age
* Newly Diagnosed Dyslipidemia Patients Including: 1) Intermediate Risk (>2 Risk Factors) With Total Cholesterol level above 200 mg/dL Or Low Density Lipoprotein-C (LDL-C) level> 130 mg/dLwho failed a 3-Month diet control period, or 2) High Risk Patients with history of Coronary artery disease Or diabetes and having a total Cholesterol> 200 mg/dL Or LDL-C level> 130 mg/dL
* Willing To Follow An National Cholesterol Education Program (NCEP) Therapeutic Lifestyle Changes (TLC) Or Similar Cholesterol-Lowering Diet For The Duration Of The Study
* Female Patients Receiving Hormone Therapy (Including Hormone Replacement Therapy, And Estrogen Antagonist/Agonist, Or Oral Contraceptives) If Maintained On A Stable Dose And Regimen For At Least 8 Weeks Prior To Visit 1 And If Willing To Continue The Same Regimen Throughout The Study

Exclusion Criteria:

* Women Who Are Pregnant Or Lactating
* Has A History Of Cancer Within The Past 5 Years (Except For Dermatological Basal Cell Or Squamous Cell Carcinoma)
* Patients Hypersensitive To Simvastatin Or Ezetimibe
* Any Condition Or Situation Which, In The Opinion Of The Investigator, Might Pose A Risk To The Patient Or Confound The Results Of The Study
* History Of Mental Instability, Drug/Alcohol Abuse Within The Past 5 Years, Or Major Psychiatric Illness Not Adequately Controlled By Pharmacotherapy
* Nephritic Syndrome Or Other Clinically Significant Renal Disease Resulting In Impaired Renal Function, Defined As Serum Creatinine ≧ 1.5 Mg/Dl
* Alanine Aminotransferase (ALT), And Aspartate Aminotransferase (AST) above 1.5 X Upper Limit Of Normal (Uln) Or With Active Liver Disease
* Congestive Heart Failure (New York Heart Association (NYHA) III Or IV), Uncontrolled Cardiac Arrythmias, Uncontrolled Hypertension (Systolic Blood Pressure (SBP) >160 mm Hg Or Diastolic Blood Pressure (DBP) >100 mm Hg), Unstable Angina Pectoris Or Severe Peripheral Artery Disease, Or Experienced Myocardial Infarction, Coronary Artery Bypass Surgery, Angioplasty Within 3 Months
* Unstable Diabetes Mellitus Patient (Hemoglobin A1c (HbA1c) > 8.5%) Or Newly Diagnosed (Within 3 Months) Or A Change In Anti-Diabetic Pharmacotherapy Within 3 Months Of Screening
* Secondary Dyslipidemia (E.G., Hypothyroidism)
* Disorders Of The Hematologic, Digestive, Or Central Nervous Systems Including Cerebrovascular Disease And Degenerative Disease That Would Limit Study Evaluation Or Participation
* History Of Active Or Chronic Hepatobiliary Disease Or Cholelithiasis But Have Not Undergone Cholecystectomy

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2007-08-01 (Actual); Primary Completion 2009-07-01 (Actual); Study Completion 2009-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang JC, Lee TY, Liou MJ, Lin CM, Pei D, Chen ZC, Liu RT, Kwok CF. Begin with the real-world patients of non-goal-achieved hypercholesterolemia in taiwan through the ezetimibe/simvastatin tablet - The BRAVO Study. Curr Med Res Opin. 2011 Aug;27(8):1645-51. doi: 10.1185/03007995.2011.594425. Epub 2011 Jun 23. PMID 21699369

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited between August 2007 and July 2009.
  In one site, 60 patients among the total 152 study population entered into the 6-week extension period after completing the base period for longer follow-up as per IRB requirement in that site.
Groups:
- Ezetimibe/Simvastatin 10/20 mg: Ezetimibe/Simvastatin 10/20 mg tablet, once daily for the 6-week period
Period: 6-week Active Treatment Period
Arm/Group | Ezetimibe/Simvastatin 10/20 mg
Started | 173
Completed | 152
Not Completed | 21
Not completed — Adverse Event | 9
Not completed — Lost to Follow-up | 10
Not completed — Transferred to branch hospital | 1
Not completed — Out of window period | 1
Period: 6 -Week Extension Period (Single Site)
Arm/Group | Ezetimibe/Simvastatin 10/20 mg
Started | 60 (Subjects who completed the first 6-week period and participated in the second 6-week study period.)
Completed | 55
Not Completed | 5
Not completed — Adverse Event | 4
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ezetimibe/Simvastatin 10/20 mg
Number analyzed (Participants) | 173
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.9 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100
  Male | 73
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 25.5 (3.4)
Baseline value of Low Density Lipoprotein-C [Mean (Standard Deviation); unit: mg/dL] | 156.8 (30.8)
Baseline value of Total Cholesterol [Mean (Standard Deviation); unit: mg/dL] | 243.7 (43.9)
Baseline value of High Density Lipoprotein-C [Mean (Standard Deviation); unit: mg/dL] | 47.1 (11.4)
Baseline value of Triglycerides [Median (Full Range); unit: mg/dL] | 145 [89 to 206]
Sitting Diastolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] | 78.5 (10.2)
Sitting Systolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] | 133.3 (16.6)

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Participants Achieving Low Density Lipoprotein-C (LDL-C) Treatment Goal After 6-week Treatment.
Description: Goal attainment percentage of LDL-C after 6-week treatment. LDL-C goal attainment was based on National Cholesterol Education program (NCEP) Adult Treatment Panel (ATP) III guidelines (2004). Newly Diagnosed Dyslipidemia Patients Including: 1)Intermediate Risk (>2 Risk Factors) with Total Cholesterol above 200 mg/dL or Low Density Lipoprotein C (LDL-C) level >130 who failed a 3-month diet control period, or 2) high risk patients with a history of coronary artery disease or diabetes having a total cholesterol >200 mg/dl or LDL-C level >130 mg/dl.
Time Frame: Baseline and week 6
Population: Intention-To-Treat (ITT) approach which included all participants who have baseline measurement, have taken at least one dose of the study drug, and have at least one post-baseline measurement.
Measure: Number; unit: Percentage of participants
Arm/Group | Ezetimibe/Simvastatin 10/20 mg
Number analyzed (Participants) | 115
Percentage of participants | 90.4

2. Primary Outcome: The Percentage of Participants Achieving Low Density Lipoprotein-C (LDL-C) Treatment Goal After 12-week Treatment.
Description: Goal attainment percentage of LDL-C after 12-week treatment. LDL-C goal attainment was based on National Cholesterol Education program (NCEP) Adult Treatment Panel (ATP) III guidelines (2004). Newly Diagnosed Dyslipidemia Patients Including: 1)Intermediate Risk (>2 Risk Factors) with Total Cholesterol above 200 mg/dL or Low Density Lipoprotein C (LDL-C) level >130 who failed a 3-month diet control period, or 2) high risk patients with a history of coronary artery disease or diabetes having a total cholesterol >200 mg/dl or LDL-C level >130 mg/dl.
Time Frame: Baseline and week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Ezetimibe/Simvastatin 10/20 mg
Number analyzed (Participants) | 49
Percentage of participants | 87.8

3. Secondary Outcome: Mean Percent Change From Baseline of Low Density Lipoprotein-Cholesterol (LDL-C) at Week 6
Time Frame: Baseline and week 6
Population: Intention-To-Treat(ITT) approach which included all participants who have baseline measurement, have taken at least one dose of the study drug, and have at least one post-baseline measurement
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Ezetimibe/Simvastatin 10/20 mg
Number analyzed (Participants) | 152
Percent Change | -51.4 (15.6)

4. Secondary Outcome: Mean Percent Change From Baseline of Total-Cholesterol (TC) at Week 6
Time Frame: Baseline and week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Ezetimibe/Simvastatin 10/20 mg
Number analyzed (Participants) | 152
Percent Change | -38.1 (11.3)

5. Secondary Outcome: Mean Percent Change From Baseline of High Density Lipoprotein-C (HDL-C) at Week 6
Time Frame: Baseline and week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Ezetimibe/Simvastatin 10/20 mg
Number analyzed (Participants) | 152
Percent Change | 4.5 (15.8)

6. Secondary Outcome: Mean Percent Change of Triglycerides From Baseline at Week 6
Time Frame: Baseline and week 6
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | Ezetimibe/Simvastatin 10/20 mg
Number analyzed (Participants) | 152
Percent Change | -22.2 [-43.6 to 0]

7. Other Pre Specified Outcome: Mean Change From Baseline of Low Density Lipoprotein-Cholesterol (LDL-C) at Week 6
Time Frame: Baseline and week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Ezetimibe/Simvastatin 10/20 mg
Number analyzed (Participants) | 152
mg/dL | -82.0 (30.8)

8. Secondary Outcome: Mean Percent Change From Baseline of Low Density Lipoprotein-Cholesterol (LDL-C) at Week 12
Time Frame: Baseline and week 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Ezetimibe/Simvastatin 10/20 mg
Number analyzed (Participants) | 55
Percent Change | -53.8 (16.7)

9. Secondary Outcome: Mean Percent Change From Baseline of Total-Cholesterol (TC) at Week 12
Time Frame: Baseline and week 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Ezetimibe/Simvastatin 10/20 mg
Number analyzed (Participants) | 55
Percent Change | -39.5 (12.2)

10. Secondary Outcome: Mean Percent Change From Baseline of High Density Lipoprotein-C (HDL-C) at Week 12
Time Frame: Baseline and week 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Ezetimibe/Simvastatin 10/20 mg
Number analyzed (Participants) | 55
Percent Change | 9.4 (20.5)

11. Secondary Outcome: Mean Percent Change of Triglycerides From Baseline at Week 12
Time Frame: Baseline and week 12
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | Ezetimibe/Simvastatin 10/20 mg
Number analyzed (Participants) | 55
Percent Change | -24.7 [-42.9 to -3.6]

12. Other Pre Specified Outcome: Mean Change From Baseline of Low Density Lipoprotein-Cholesterol (LDL-C) at Week 12
Time Frame: Baseline and week 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Ezetimibe/Simvastatin 10/20 mg
Number analyzed (Participants) | 55
mg/dL | -85.6 (31.7)

ADVERSE EVENTS:
Arm/Group | Ezetimibe/Simvastatin 10/20 mg
Serious Adverse Events (participants affected / at risk) | 1/173
Other Adverse Events (participants affected / at risk) | 34/173
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ezetimibe/Simvastatin 10/20 mg (N=173)
Peptic Ulcer (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ezetimibe/Simvastatin 10/20 mg (N=173)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (7)
Dizziness (Nervous system disorders) | 5 (5)
Flatulence (Gastrointestinal disorders) | 2 (2)
Upper Respiratory Infection (Infections and infestations) | 7 (7)
Increased Creatine Phosphokinase (CPK) (Investigations) | 6 (6)
Increased Serum Glutamic Pyruvic Transaminase (SGPT) (Investigations) | 5 (5)
Fatigue (General disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.